CLINICAL TRIAL: NCT01077622
Title: A Phase I/II, a Single Arm, Open-label Study of Ofatumumab (GSK1841157) in Patients With Previously Treated Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 112758
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2013-10

CONDITIONS: Leukaemia, Lymphocytic, Chronic
MeSH Terms: conditions — Leukemia, B-Cell | interventions — ofatumumab

ARMS (1):
- 2000 mg dose (Experimental): ofatumumab , 300mg followed by 7 weekly infusions 2000 mg, followed by 4 monthly infusions 2000mg
  Interventions: Drug: ofatumumab 100 mg, 1000 mg / vial

INTERVENTIONS:
Drug: ofatumumab 100 mg, 1000 mg / vial — ofatumumab , 300mg followed by 7 weekly infusions 2000 mg, followed by 4 monthly infusions 2000mg

SUMMARY:
Ofatumumab is an IgG1κ fully human monoclonal antibody (mAb) that specifically recognizes an epitope on the human differentiation antigen CD20 molecule. In vitro and in vivo studies demonstrated that ofatumumab depletes CD20 positive (CD20+) B cells through complement-dependent cytotoxicity (CDC) and antibody-dependent cell-mediated cytotoxicity (ADCC), which results in the antitumour effect.

This is an open-label study to evaluate safety, tolerability, efficacy and PK profile of ofatumumab monotherapy in chronic lymphocytic leukemia (CLL) patients. Ofatumumab will be administered intravenously at the first dose of 300mg followed by 7 weekly infusions of 2000mg, followed by 4 infusions of 2000mg at every 4 weeks.

Primary objective of the study (Part A) is to evaluate tolerability, and the study (Part B) is to assess overall response rate in CLL population.

10 subjects will be enrolled into this study. Subjects will be followed for 48 weeks.

DETAILED DESCRIPTION:
Ofatumumab is an IgG1κ fully human monoclonal antibody (mAb) that specifically recognizes an epitope on the human differentiation antigen CD20 molecule. In vitro and in vivo studies demonstrated that ofatumumab depletes CD20 positive (CD20+) B cells through complement-dependent cytotoxicity (CDC) and antibody-dependent cell-mediated cytotoxicity (ADCC), which results in the antitumour effect.

This is an open-label study to evaluate safety, tolerability, efficacy and PK profile of ofatumumab monotherapy in chronic lymphocytic leukemia (CLL) patients. Ofatumumab will be administered intravenously at the first dose of 300mg followed by 7 weekly infusions of 2000mg, followed by 4 infusions of 2000mg at every 4 weeks.

Primary objective of the study (Part A) is to evaluate tolerability, and the study (Part B) is to assess overall response rate in CLL population.

10 subjects will be enrolled into this study. Subjects will be followed for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria at the time of screening:

* Patients who gave consent to this study participation and signed into informed consent form.
* Previously treated(Patients who received at least one prior CLL therapy and have either relapsed or have refractory disease, both requiring therapy.) CLL with at least 5 x 109 B lymphocytes/ L (5000/μL). The diagnosis of CLL requires CD5, CD19, CD20 and CD23 positivity, according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) guidelines [Hallek, 2008].
* Laboratory test values meet the following criteria which indicate that patients have sufficient physiological functions;

Neutrophils:1≥ 500 /mm3 ALT ≤ 2.5 times upper local normal limit Creatinine ≤ 1.5 times upper local normal limit Total bilirubin≤ 1.5 times upper local normal limit

1:Patients should not receive any hematopoietic cytokine such as G-CSF preparations within 1 week before screening laboratory test for neutrophil counting.

- Patients who passed the following periods from the last anti-cancer treatments at the time of screening: At least 4 weeks after anti-cancer chemotherapy. At least 4 weeks after anti-cancer radiotherapy. At least 4 weeks after glucocorticoids treatment for CLL unless ≤ 10 mg of prednisolone /day.

At least 12 weeks after radio-immunotherapy and/or antibody therapy.

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1, or 2.
* Life expectancy more than 24 weeks after screening test.
* Aged ≥ 20 (at the time of signing informed consent).
* Patients possible to stay at the trial site for at least two days (the day of the first infusion and a subsequent day).

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria is met:

* Active malignancy which needs therapy with anti-cancer drug, except for CLL.
* Known Richter's transformation.
* Previous autologous stem cell transplantation, within 24 weeks prior to screening.
* Previous allogenic stem cell transplantation.
* Known CNS involvement.
* History of significant cerebrovascular disease.
* Current cardiac disease requiring medical treatment (e.g. atrial flutter treated with acetylsalicylic acid and beta blocking agents).
* Chronic or active infectious disease requiring systemic (intravenous or oral) treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis and tuberculosis.
* Suspected/known immediate or delayed hypersensitivity to components of ofatumumab.
* Patients previously treated with ofatumumab.
* Positive serology test for any of HBsAg, anti-HBcAb or anti-HCVAb. If only anti-HBcAb results is positive, HBV-DNA test will be performed. If HBV-DNA results in negative, the patient is eligible.
* HIV positivity.
* Pregnant or lactating women.
* Women of childbearing potential not willing to use adequate contraception during the study and one year after the last dose of ofatumumab, and male patients not willing to use adequate contraception during the study. Adequate contraception is defined as follows but not limited to; Abstinence. Oral Contraceptive (exclude oral progesterone alone). Intrauterine device (IUD) or intrauterine system (IUS). Male partner sterilization. Double barrier method: condom or occlusive cap (diaphragm or cervical / vault caps) plus spermicidal agent (gel / film) etc.
* Use of an investigational drug within 4 weeks prior to screening.
* Current participation in any other clinical study.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease.
* Patients who an investigator (or sub investigator) judges ineligible to this study.

Note; Child-bearing potential: a woman with functioning ovaries and uterine, or no documented sterility (i.e., a woman with functioning ovaries who have a current documented tubal ligation, women who have had a hysterectomy, women who are post-menopausal, or women who have had both ovaries surgically removed).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09-01; Primary Completion 2011-04-01 (Actual); Study Completion 2011-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Japan (4):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab: Participants received intravenous ofatumumab at an initial dose of 300 milligrams (mg). One week after the initial dose, participants received 7 infusions of 2000 mg at weekly intervals. Five weeks after the last 2000 mg infusion, participants received 4 infusions of 2000 mg at 4-week intervals.
Period: Overall Study
Arm/Group | Ofatumumab
Started | 10
Completed | 7
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Asian - East Asian Heritage | 1
  Asian - Japanese Heritage | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A DLT was defined as the following toxicological findings, according to the Common Terminology Criteria for Adverse Events (AE) v3.0: any treatment-related Grade (G) >=3 non-hematotoxic AE, occurrence of G3 infusion reaction (treatment-related AE) at the day of infusion in a participant who received pre-medication or appropriate management during infusion (glucocorticoid) (the severity of the AE must have remained as >= G3 until the next day); and any of following: >= G4 hematotoxic treatment-related AEs (neutropenia lasting 7 days or more, febrile neutropenia).
Time Frame: Up to Week 8
Population: All Subjects Population: all participants who received at least one dose of investigational drug. The first 3 participants enrolled in the study were evaluated for DLT according to study design.
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 3
participants | 0

2. Primary Outcome: Percentage of Participants (Par.) With Objective Response (OR), Defined as Complete Remission (CR), CR Incomplete (CRi), Partial Remission (PR), and Nodular PR (nPR) as Assessed by a Safety and Evaluation Review Committee (SERC) and the Investigator
Description: Par. were evaluated in accordance with the National Cancer Institute-sponsored Working Group. CR: no lymphadenopathy (Ly)/hepatomegaly/splenomegaly/constitutional symptoms; neutrophils >=1.5*10^9/liter (L), platelets >100*10^9/L, hemoglobin >11.0 grams/deciliter, lymphocytes (LC) <4.0*10^9/L, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to chronic lymphocytic leukemia but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen, etc. nPR: nodules in BM.
Time Frame: Up to Week 48
Population: All Subjects Population
Measure: Number; unit: Percentage of participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
Percentage of participants
  SERC | 70
  Investigator | 70
Statistical Analysis 1: Comparison: Ofatumumab; Test type: Superiority or Other; percentage of participants = 70, 95% CI 2-sided [34.8 to 93.3] — SERC assessment
Statistical Analysis 2: Comparison: Ofatumumab; Test type: Superiority or Other; percentage of participants = 70, 95% CI 2-sided [34.8 to 93.3] — Investigator assessment

3. Secondary Outcome: Progression-free Survival (PFS) as Assessed by a SERC
Description: PFS is defined as the time from the start of treatment to the first documented sign of progressive disease (PD) or death due to any cause (whichever occurs earlier).
Time Frame: Up to Week 48
Population: All Subjects Population: only those participants who progressed or died during the study were evaluated.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab
Number analyzed (Participants) | 2
Weeks | NA [36.1 to NA] — Because the number of evaluable participants is small (2/10), it is not possible to estimate the median value and the upper limit of the 95% confidence interval of the median value for PFS.

4. Secondary Outcome: Duration of Response as Assessed by a SERC
Description: Duration of response is defined as the time from the first documented evidence of PR or better until the first documented sign of PD or death due to any reason in participants with PR or better.
Time Frame: Up to Week 48
Population: All Subjects Population: only those participants classified as responders for the assessment of objective response were evaluated.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab
Number analyzed (Participants) | 7
Weeks | NA [NA to NA] — None of the seven responders progressed at the time of the analysis; thus, no data can be presented.

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the first infusion of investigational drug to death due to any cause.
Time Frame: Up to Week 48
Population: All Subjects Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
Weeks | NA [NA to NA] — All 10 participants were alive at the time of last follow-up.

6. Secondary Outcome: Time to Response as Assessed by a SERC
Description: Time to response is defined as the time from the first infusion of investigational drug to the first response (PR or better).
Time Frame: Up to Week 48
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab
Number analyzed (Participants) | 7
Weeks | 8.1 [8.0 to 24.1]

7. Secondary Outcome: Time to Next Chronic Lymphocytic Leukemia (CLL) Therapy as Assessed by a SERC
Description: Time to next CLL therapy is defined as the time from the first infusion of investigational drug to the first administration of the next CLL treatment. CLL therapy includes anti-cancer chemotherapy, anti-cancer radiotherapy, radio-immunotherapy, and antibody therapy.
Time Frame: Up to Week 48
Population: All Subjects Population: only those participants who received CLL therapy were evaluated.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab
Number analyzed (Participants) | 2
Weeks | NA [NA to NA] — Because the number of evaluable participants is small (2/10), it is not possible to calculate the median value for time to next CLL therapy.

8. Secondary Outcome: Mean Laboratory Data for Hemoglobin at the Indicated Weeks as Assessed by the Investigator
Description: Blood samples of the participants were collected for the assessment of hemoglobin.
Time Frame: Day 1; Weeks 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 28, 36, and 48
Population: All Subjects Population. Only participants remaining in the study and contributing evaluable data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
Grams per liter (g/L)
  Day 1, n=10 | 115.7 (15.44)
  Week 1, n=10 | 116.0 (15.46)
  Week 2, n=10 | 117.4 (16.37)
  Week 3, n=10 | 117.0 (18.68)
  Week 4, n=10 | 116.1 (18.53)
  Week 5, n=10 | 116.4 (17.83)
  Week 6, n=10 | 118.1 (16.25)
  Week 7, n=10 | 118.4 (20.06)
  Week 8, n=10 | 119.8 (20.35)
  Week 12, n=10 | 122.6 (20.55)
  Week 16, n=10 | 125.6 (21.08)
  Week 20, n=10 | 127.8 (21.81)
  Week 24, n=10 | 127.8 (22.31)
  Week 28, n=9 | 126.2 (21.49)
  Week 36, n=9 | 128.1 (20.91)
  Week 48, n=7 | 137.1 (11.01)

9. Secondary Outcome: Mean Laboratory Data for Lymphocytes at the Indicated Weeks as Assessed by the Investigator
Description: Blood samples of the participants were collected for the assessment of lymphocytes.
Time Frame: Day 1; Weeks 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Giga (10^9) per liter (GI/L)
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
Giga (10^9) per liter (GI/L)
  Day 1, n=10 | 42.6038 (41.66244)
  Week 1, n=10 | 29.6861 (33.19072)
  Week 2, n=10 | 8.2290 (6.76264)
  Week 3, n=10 | 6.9065 (6.81649)
  Week 4, n=10 | 4.0446 (2.70652)
  Week 5, n=10 | 2.9535 (1.47227)
  Week 6, n=10 | 2.8063 (1.43681)
  Week 7, n=10 | 2.4792 (1.20853)
  Week 8, n=10 | 2.1515 (0.94237)
  Week 12, n=10 | 1.8058 (0.95653)
  Week 16, n=10 | 1.9575 (1.09880)
  Week 20, n=10 | 1.8388 (1.22494)
  Week 24, n=10 | 1.8500 (1.33979)
  Week 28, n=9 | 1.6405 (1.05653)
  Week 36, n=9 | 3.5754 (5.38456)
  Week 48, n=7 | 1.5099 (0.72285)

10. Secondary Outcome: Mean Laboratory Data for Lymphocytes as a Percentage in the Bone Marrow at the Indicated Weeks as Assessed by the Investigator
Description: Bone marrow (BM) aspiration was performed, and the bone marrow smears were prepared for the assessment of lymphocytes in the BM.
Time Frame: Weeks 8, 16, 24, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes in the BM
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
Percentage of lymphocytes in the BM
  Week 8, n=8 | 57.90 (23.492)
  Week 16, n=5 | 38.04 (14.647)
  Week 24, n=7 | 36.96 (14.961)
  Week 36, n=6 | 30.00 (17.030)
  Week 48, n=5 | 23.26 (9.651)

11. Secondary Outcome: Mean Laboratory Data for Total Neutrophils (Total Absolute Neutrophil Count [ANC]) at the Indicated Weeks as Assessed by the Investigator
Description: Blood samples of the participants were collected for the assessment of total neutrophils.
Time Frame: Day 1; Weeks 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
GI/L
  Day 1, n=10 | 4.3103 (1.91880)
  Week 1, n=10 | 3.9316 (2.37732)
  Week 2, n=10 | 3.2158 (1.62185)
  Week 3, n=10 | 2.7873 (1.16531)
  Week 4, n=10 | 2.4570 (1.22611)
  Week 5, n=10 | 2.3908 (0.99250)
  Week 6, n=10 | 2.1747 (1.00743)
  Week 7, n=10 | 2.1612 (1.22393)
  Week 8, n=10 | 2.2136 (1.22993)
  Week 12, n=10 | 1.9814 (0.90783)
  Week 16, n=10 | 1.9915 (1.00746)
  Week 20, n=10 | 2.2165 (1.29881)
  Week 24, n=10 | 2.3093 (1.18840)
  Week 28, n=9 | 2.2069 (1.57995)
  Week 36, n=9 | 2.3482 (1.04228)
  Week 48, n=7 | 3.0431 (1.67580)

12. Secondary Outcome: Mean Laboratory Data for Platelet Count at the Indicated Weeks as Assessed by the Investigator
Description: Blood samples of the participants were collected for the assessment of platelets.
Time Frame: Day 1; Weeks 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
GI/L
  Day 1, n=10 | 106.5 (31.69)
  Week 1, n=10 | 104.0 (45.45)
  Week 2, n=10 | 100.1 (37.21)
  Week 3, n=10 | 118.3 (40.90)
  Week 4, n=10 | 114.9 (46.26)
  Week 5, n=10 | 111.5 (47.11)
  Week 6, n=10 | 115.7 (49.86)
  Week 7, n=10 | 121.4 (54.65)
  Week 8, n=10 | 127.7 (64.44)
  Week 12, n=10 | 120.1 (46.29)
  Week 16, n=10 | 124.3 (46.00)
  Week 20, n=10 | 134.0 (41.66)
  Week 24, n=10 | 136.6 (44.14)
  Week 28, n=9 | 128.9 (41.64)
  Week 36, n=9 | 143.0 (43.19)
  Week 48, n=7 | 130.7 (53.70)

13. Secondary Outcome: Percentage of Bone Marrow Infiltration at the Indicated Weeks as Assessed by a SERC
Description: SERC assessed bone marrow infiltration with the bone marrow smears of participants provided by trial sites.
Time Frame: Weeks 8, 16, 24, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of bone marrow infiltration
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
Percentage of bone marrow infiltration
  Week 8, n=8 | 57.90 (23.492)
  Week 16, n=5 | 38.04 (14.647)
  Week 24, n=7 | 36.96 (14.961)
  Week 36, n=6 | 29.13 (17.379)
  Week 48, n=5 | 23.26 (9.651)

14. Secondary Outcome: Mean Laboratory Data for Lymphocytes at the Indicated Weeks as Assessed by a SERC
Description: SERC assessed lymphocytes based on the data provided by trial sites.
Time Frame: Weeks 8, 16, 24, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
GI/L
  Week 8, n=8 | 2.0120 (1.03095)
  Week 16, n=6 | 1.7975 (1.05163)
  Week 24, n=7 | 1.8784 (1.56286)
  Week 36, n=6 | 2.1213 (2.65560)
  Week 48, n=5 | 1.6284 (0.70741)

15. Secondary Outcome: Mean Laboratory Data for Lymphocytes as a Percentage in the Bone Marrow at the Indicated Weeks as Assessed by a SERC
Description: SERC assessed lymphocytes in the bone marrow (BM) based on the data with BM smears provided by trial sites.
Time Frame: Weeks 8, 16, 24, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes in BM
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
percentage of lymphocytes in BM
  Week 8, n=8 | 57.90 (23.492)
  Week 16, n=5 | 38.04 (14.647)
  Week 24, n=7 | 36.96 (14.961)
  Week 36, n=6 | 29.13 (17.379)
  Week 48, n=5 | 23.26 (9.651)

16. Secondary Outcome: Mean Laboratory Data for Total Neutrophils (Total ANC) at the Indicated Weeks as Assessed by a SERC
Description: SERC assessed total neutrophils based on the data provided by trial sites.
Time Frame: Weeks 8, 16, 24, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
GI/L
  Week 8, n=8 | 2.3159 (1.35507)
  Week 16, n=6 | 2.5803 (1.04075)
  Week 24, n=7 | 2.8706 (1.39803)
  Week 36, n=6 | 2.1957 (0.89898)
  Week 48, n=5 | 2.6242 (1.05912)

17. Secondary Outcome: Number of Peripheral Blood Cluster of Differentiation (CD) CD19+ CD20+ Cells
Description: CD19+ CD20+ cells in the peripheral blood were counted as measures of malignant B-cells and were measured by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus.
Time Frame: Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
GI/L
  Day 1, n=10 | 33.1140 (39.40966)
  Week 1, n=9 | 19.6438 (35.81756)
  Week 2, n=10 | 0.0060 (0.01151)
  Week 4, n=10 | 0.0565 (0.16699)
  Week 6, n=10 | 0.0022 (0.00258)
  Week 8, n=9 | 0.0006 (0.00136)
  Week 12, n=10 | 0.0006 (0.00116)
  Week 16, n=10 | 0.0003 (0.00058)
  Week 20, n=10 | 0.0005 (0.00087)
  Week 24, n=10 | 0.0002 (0.00037)
  Week 28, n=9 | 0.0003 (0.00093)
  Week 36, n=8 | 0.2525 (0.71266)
  Week 48, n=7 | 0.0914 (0.10259)

18. Secondary Outcome: Number of Peripheral Blood CD20+ CD23+ Cells
Description: CD20+ CD23+ cells in the peripheral blood were counted as measures of malignant B-cells and were measured by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus.
Time Frame: Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
GI/L
  Day 1, n=10 | 19.9791 (27.06441)
  Week 1, n=9 | 8.9466 (21.59662)
  Week 2, n=10 | 0.0319 (0.04010)
  Week 4, n=10 | 0.0685 (0.14483)
  Week 6, n=10 | 0.0099 (0.01869)
  Week 8, n=9 | 0.0047 (0.01131)
  Week 12, n=10 | 0.0080 (0.02270)
  Week 16, n=10 | 0.0111 (0.03162)
  Week 20, n=10 | 0.0048 (0.01277)
  Week 24, n=10 | 0.0057 (0.01553)
  Week 28, n=9 | 0.0002 (0.00040)
  Week 36, n=8 | 0.2147 (0.60466)
  Week 48, n=7 | 0.0773 (0.09355)

19. Secondary Outcome: Number of Peripheral Blood CD19+ CD23+ Cells
Description: CD19+ CD23+ cells in the peripheral blood were counted as measures of malignant B-cells and were measured by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus.
Time Frame: Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
GI/L
  Day 1, n=10 | 23.8046 (28.66936)
  Week 1, n=9 | 17.4769 (22.30923)
  Week 2, n=10 | 4.6972 (6.14672)
  Week 4, n=10 | 1.8230 (2.49206)
  Week 6, n=10 | 0.4858 (0.55687)
  Week 8, n=9 | 0.2252 (0.25765)
  Week 12, n=10 | 0.2122 (0.26787)
  Week 16, n=10 | 0.1961 (0.34108)
  Week 20, n=10 | 0.1464 (0.33132)
  Week 24, n=10 | 0.1330 (0.23961)
  Week 28, n=9 | 0.1123 (0.26130)
  Week 36, n=8 | 0.2687 (0.71524)
  Week 48, n=7 | 0.0886 (0.11398)

20. Secondary Outcome: Number of Peripheral Blood CD19+ CD5+ Cells
Description: CD19+ CD5+ cells in the peripheral blood were counted as measures of malignant B-cells and were measured by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus.
Time Frame: Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
GI/L
  Day 1, n=10 | 36.0022 (36.64910)
  Week 1, n=9 | 27.9129 (32.61649)
  Week 2, n=10 | 5.4212 (6.55286)
  Week 4, n=10 | 2.2158 (2.62609)
  Week 6, n=10 | 0.5799 (0.63484)
  Week 8, n=9 | 0.2338 (0.27058)
  Week 12, n=10 | 0.2420 (0.32493)
  Week 16, n=10 | 0.2425 (0.38048)
  Week 20, n=10 | 0.1943 (0.38386)
  Week 24, n=10 | 0.1719 (0.29401)
  Week 28, n=9 | 0.1449 (0.25617)
  Week 36, n=8 | 0.2858 (0.73543)
  Week 48, n=7 | 0.1200 (0.14511)

21. Secondary Outcome: Number of Peripheral Blood CD20+ CD5+ Cells
Description: CD20+ CD5+ cells in the peripheral blood were counted as measures of malignant B-cells and were measured by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus.
Time Frame: Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
GI/L
  Day 1, n=10 | 32.9606 (39.50102)
  Week 1, n=9 | 19.3999 (35.56146)
  Week 2, n=10 | 0.0134 (0.01696)
  Week 4, n=10 | 0.0493 (0.13576)
  Week 6, n=10 | 0.0024 (0.00185)
  Week 8, n=9 | 0.0029 (0.00136)
  Week 12, n=10 | 0.0020 (0.00160)
  Week 16, n=10 | 0.0062 (0.00907)
  Week 20, n=10 | 0.0026 (0.00147)
  Week 24, n=10 | 0.0036 (0.00258)
  Week 28, n=9 | 0.0022 (0.00214)
  Week 36, n=8 | 0.2597 (0.72781)
  Week 48, n=7 | 0.0968 (0.11682)

22. Secondary Outcome: Number of Peripheral Blood CD23+ CD5+ Cells
Description: CD23+ CD5+ cells in the peripheral blood were counted as measures of malignant B-cells and were measured by flow cytometry. Flow cytometry is a technique for counting and examining microscopic particles with an electronic detection apparatus.
Time Frame: Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
GI/L
  Day 1, n=10 | 22.7190 (25.17338)
  Week 1, n=9 | 17.2018 (21.23454)
  Week 2, n=10 | 4.5264 (6.03353)
  Week 4, n=10 | 1.8255 (2.49671)
  Week 6, n=10 | 0.4714 (0.50306)
  Week 8, n=9 | 0.2095 (0.23907)
  Week 12, n=10 | 0.2114 (0.27306)
  Week 16, n=10 | 0.1866 (0.34514)
  Week 20, n=10 | 0.1478 (0.32088)
  Week 24, n=10 | 0.1327 (0.23698)
  Week 28, n=9 | 0.1035 (0.23789)
  Week 36, n=8 | 0.2570 (0.68983)
  Week 48, n=7 | 0.1062 (0.13388)

23. Secondary Outcome: Ratio of Immunoglobulin (Ig) Kappa/Ig Lambda
Description: Peripheral blood Ig kappa and Ig lambda were measured using flow cytometry. Abnormality of a ratio of Ig kappa and Ig lambda indicates clonality of lymphocytes. A normal range of this parameter is between 1.0 and 3.2.
Time Frame: Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Ratio of Ig kappa/Ig lambda
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
Ratio of Ig kappa/Ig lambda
  Day 1, n=10 | 34.710 (38.2375)
  Week 1, n=9 | 36.604 (36.9383)
  Week 2, n=10 | 15.928 (26.5203)
  Week 4, n=10 | 9.451 (25.1555)
  Week 6, n=10 | 7.263 (20.3014)
  Week 8, n=9 | 6.427 (16.7389)
  Week 12, n=10 | 3.799 (8.8774)
  Week 16, n=10 | 2.150 (3.8972)
  Week 20, n=10 | 2.017 (3.8733)
  Week 24, n=10 | 1.608 (2.6223)
  Week 28, n=9 | 1.647 (2.3965)
  Week 36, n=8 | 1.693 (1.8636)
  Week 48, n=7 | 3.368 (5.2575)

24. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline (BL) in Night Sweats at the Indicated Weeks
Description: Night sweats are one of the clinical characteristics of CLL. B symptoms are systemic symptoms of fever, night sweats, weight loss, and extreme fatigue, which can be associated with CLL. Participants who had night sweats at BL, and still had night sweats at Week 1, for example, are represented in the BL, yes; Week 1, yes category. Participants who had night sweats at BL, but did not have night sweats at Week 1 are represented in the BL, yes; Week 1, no category.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
participants
  BL, yes; Week 1, yes; n=10 | 1
  BL, yes; Week 1, no; n=10 | 0
  BL, no; Week 1, yes; n=10 | 0
  BL, no; Week 1, no; n=10 | 9
  BL, yes; Week 2, yes; n=10 | 1
  BL, yes; Week 2, no; n=10 | 0
  BL, no; Week 2, yes; n=10 | 0
  BL, no; Week 2, no; n=10 | 9
  BL, yes; Week 3, yes; n=10 | 1
  BL, yes; Week 3, no; n=10 | 0
  BL, no; Week 3, yes; n=10 | 0
  BL, no; Week 3, no; n=10 | 9
  BL, yes; Week 4, yes; n=10 | 1
  BL, yes; Week 4, no; n=10 | 0
  BL, no; Week 4, yes; n=10 | 0
  BL, no; Week 4, no; n=10 | 9
  BL, yes; Week 5, yes; n=10 | 0
  BL, yes; Week 5, no; n=10 | 0
  BL, no; Week 5, yes; n=10 | 1
  BL, no; Week 5, no; n=10 | 9
  BL, yes; Week 6, yes; n=10 | 0
  BL, yes; Week 6, no; n=10 | 0
  BL, no; Week 6, yes; n=10 | 1
  BL, no; Week 6, no; n=10 | 9
  BL, yes; Week 7, yes; n=10 | 0
  BL, yes; Week 7, no; n=10 | 0
  BL, no; Week 7, yes; n=10 | 1
  BL, no; Week 7, no; n=10 | 9
  BL, yes; Week 8, yes; n=10 | 0
  BL, yes; Week 8, no; n=10 | 0
  BL, no; Week 8, yes; n=10 | 1
  BL, no; Week 8, no; n=10 | 9
  BL, yes; Week 12, yes; n=10 | 0
  BL, yes; Week 12, no; n=10 | 0
  BL, no; Week 12, yes; n=10 | 1
  BL, no; Week 12, no; n=10 | 9
  BL, yes; Week 16, yes; n=10 | 0
  BL, yes; Week 16, no; n=10 | 0
  BL, no; Week 16, yes; n=10 | 1
  BL, no; Week 16, no; n=10 | 9
  BL, yes; Week 20, yes; n=10 | 0
  BL, yes; Week 20, no; n=10 | 0
  BL, no; Week 20, yes; n=10 | 1
  BL, no; Week 20, no; n=10 | 9
  BL, yes; Week 24, yes; n=10 | 0
  BL, yes; Week 24, no; n=10 | 0
  BL, no; Week 24, yes; n=10 | 1
  BL, no; Week 24, no; n=10 | 9
  BL, yes; Week 28, yes; n=9 | 0
  BL, yes; Week 28, no; n=9 | 0
  BL, no; Week 28, yes; n=9 | 1
  BL, no; Week 28, no; n=9 | 8
  BL, yes; Week 36, yes; n=9 | 0
  BL, yes; Week 36, no; n=9 | 0
  BL, no; Week 36, yes; n=9 | 1
  BL, no; Week 36, no; n=9 | 8
  BL, yes; Week 48, yes; n=7 | 0
  BL, yes; Week 48, no; n=7 | 0
  BL, no; Week 48, yes; n=7 | 0
  BL, no; Week 48, no; n=7 | 7

25. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline (BL) in Weight Loss at the Indicated Weeks
Description: Weight loss is one of the clinical characteristics of CLL. B symptoms are systemic symptoms of fever, night sweats, weight loss, and extreme fatigue, which can be associated with CLL. Participants who had weight loss at BL, and still had weight loss at Week 1, for example, are represented in the BL, yes; Week 1, yes category. Participants who had weight loss at BL, but did not have weight loss at Week 1 are represented in the BL, yes; Week 1, no category.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
participants
  BL, yes; Week 1, yes; n=10 | 0
  BL, yes; Week 1, no; n=10 | 0
  BL, no; Week 1, yes; n=10 | 0
  BL, no; Week 1, no; n=10 | 10
  BL, yes; Week 2, yes; n=10 | 0
  BL, yes; Week 2, no; n=10 | 0
  BL, no; Week 2, yes; n=10 | 0
  BL, no; Week 2, no; n=10 | 10
  BL, yes; Week 3, yes; n=10 | 0
  BL, yes; Week 3, no; n=10 | 0
  BL, no; Week 3, yes; n=10 | 0
  BL, no; Week 3, no; n=10 | 10
  BL, yes; Week 4, yes; n=10 | 0
  BL, yes; Week 4, no; n=10 | 0
  BL, no; Week 4, yes; n=10 | 0
  BL, no; Week 4, no; n=10 | 10
  BL, yes; Week 5, yes; n=10 | 0
  BL, yes; Week 5, no; n=10 | 0
  BL, no; Week 5, yes; n=10 | 0
  BL, no; Week 5, no; n=10 | 10
  BL, yes; Week 6, yes; n=10 | 0
  BL, yes; Week 6, no; n=10 | 0
  BL, no; Week 6, yes; n=10 | 0
  BL, no; Week 6, no; n=10 | 10
  BL, yes; Week 7, yes; n=10 | 0
  BL, yes; Week 7, no; n=10 | 0
  BL, no; Week 7, yes; n=10 | 0
  BL, no; Week 7, no; n=10 | 10
  BL, yes; Week 8, yes; n=10 | 0
  BL, yes; Week 8, no; n=10 | 0
  BL, no; Week 8, yes; n=10 | 0
  BL, no; Week 8, no; n=10 | 10
  BL, yes; Week 12, yes; n=10 | 0
  BL, yes; Week 12, no; n=10 | 0
  BL, no; Week 12, yes; n=10 | 0
  BL, no; Week 12, no; n=10 | 10
  BL, yes; Week 16, yes; n=10 | 0
  BL, yes; Week 16, no; n=10 | 0
  BL, no; Week 16, yes; n=10 | 0
  BL, no; Week 16, no; n=10 | 10
  BL, yes; Week 20, yes; n=10 | 0
  BL, yes; Week 20, no; n=10 | 0
  BL, no; Week 20, yes; n=10 | 0
  BL, no; Week 20, no; n=10 | 10
  BL, yes; Week 24, yes; n=10 | 0
  BL, yes; Week 24, no; n=10 | 0
  BL, no; Week 24, yes; n=10 | 0
  BL, no; Week 24, no; n=10 | 10
  BL, yes; Week 28, yes; n=9 | 0
  BL, yes; Week 28, no; n=9 | 0
  BL, no; Week 28, yes; n=9 | 0
  BL, no; Week 28, no; n=9 | 9
  BL, yes; Week 36, yes; n=9 | 0
  BL, yes; Week 36, no; n=9 | 0
  BL, no; Week 36, yes; n=9 | 0
  BL, no; Week 36, no; n=9 | 9
  BL, yes; Week 48, yes; n=7 | 0
  BL, yes; Week 48, no; n=7 | 0
  BL, no; Week 48, yes; n=7 | 0
  BL, no; Week 48, no; n=7 | 7

26. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline (BL) in Fever at the Indicated Weeks
Description: Fever is one of the clinical characteristics of CLL. B symptoms are systemic symptoms of fever, night sweats, weight loss, and extreme fatigue, which can be associated with CLL. Participants who had fever at BL, and still had fever at Week 1, for example, are represented in the BL, yes; Week 1, yes category. Participants who had fever at BL, but did not have fever at Week 1 are represented in the BL, yes; Week 1, no category.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
participants
  BL, yes; Week 1, yes; n=10 | 0
  BL, yes; Week 1, no; n=10 | 0
  BL, no; Week 1, yes; n=10 | 0
  BL, no; Week 1, no; n=10 | 10
  BL, yes; Week 2, yes; n=10 | 0
  BL, yes; Week 2, no; n=10 | 0
  BL, no; Week 2, yes; n=10 | 0
  BL, no; Week 2, no; n=10 | 10
  BL, yes; Week 3, yes; n=10 | 0
  BL, yes; Week 3, no; n=10 | 0
  BL, no; Week 3, yes; n=10 | 0
  BL, no; Week 3, no; n=10 | 10
  BL, yes; Week 4, yes; n=10 | 0
  BL, yes; Week 4, no; n=10 | 0
  BL, no; Week 4, yes; n=10 | 0
  BL, no; Week 4, no; n=10 | 10
  BL, yes; Week 5, yes; n=10 | 0
  BL, yes; Week 5, no; n=10 | 0
  BL, no; Week 5, yes; n=10 | 0
  BL, no; Week 5, no; n=10 | 10
  BL, yes; Week 6, yes; n=10 | 0
  BL, yes; Week 6, no; n=10 | 0
  BL, no; Week 6, yes; n=10 | 0
  BL, no; Week 6, no; n=10 | 10
  BL, yes; Week 7, yes; n=10 | 0
  BL, yes; Week 7, no; n=10 | 0
  BL, no; Week 7, yes; n=10 | 0
  BL, no; Week 7, no; n=10 | 10
  BL, yes; Week 8, yes; n=10 | 0
  BL, yes; Week 8, no; n=10 | 0
  BL, no; Week 8, yes; n=10 | 0
  BL, no; Week 8, no; n=10 | 10
  BL, yes; Week 12, yes; n=10 | 0
  BL, yes; Week 12, no; n=10 | 0
  BL, no; Week 12, yes; n=10 | 0
  BL, no; Week 12, no; n=10 | 10
  BL, yes; Week 16, yes; n=10 | 0
  BL, yes; Week 16, no; n=10 | 0
  BL, no; Week 16, yes; n=10 | 0
  BL, no; Week 16, no; n=10 | 10
  BL, yes; Week 20, yes; n=10 | 0
  BL, yes; Week 20, no; n=10 | 0
  BL, no; Week 20, yes; n=10 | 0
  BL, no; Week 20, no; n=10 | 10
  BL, yes; Week 24, yes; n=10 | 0
  BL, yes; Week 24, no; n=10 | 0
  BL, no; Week 24, yes; n=10 | 0
  BL, no; Week 24, no; n=10 | 10
  BL, yes; Week 28, yes; n=9 | 0
  BL, yes; Week 28, no; n=9 | 0
  BL, no; Week 28, yes; n=9 | 0
  BL, no; Week 28, no; n=9 | 9
  BL, yes; Week 36, yes; n=9 | 0
  BL, yes; Week 36, no; n=9 | 0
  BL, no; Week 36, yes; n=9 | 0
  BL, no; Week 36, no; n=9 | 9
  BL, yes; Week 48, yes; n=7 | 0
  BL, yes; Week 48, no; n=7 | 0
  BL, no; Week 48, yes; n=7 | 0
  BL, no; Week 48, no; n=7 | 7

27. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline (BL) in Extreme Fatigue at the Indicated Weeks
Description: Extreme fatigue is one of the clinical characteristics of CLL. B symptoms are systemic symptoms of fever, night sweats, weight loss, and extreme fatigue, which can be associated with CLL. Participants who had extreme fatigue at BL, and still had extreme fatigue at Week 1, for example, are represented in the BL, yes; Week 1, yes category. Participants who had extreme fatigue at BL, but did not have extreme fatigue at Week 1 are represented in the BL, yes; Week 1, no category.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
participants
  BL, yes; Week 1, yes; n=10 | 0
  BL, yes; Week 1, no; n=10 | 0
  BL, no; Week 1, yes; n=10 | 0
  BL, no; Week 1, no; n=10 | 10
  BL, yes; Week 2, yes; n=10 | 0
  BL, yes; Week 2, no; n=10 | 0
  BL, no; Week 2, yes; n=10 | 0
  BL, no; Week 2, no; n=10 | 10
  BL, yes; Week 3, yes; n=10 | 0
  BL, yes; Week 3, no; n=10 | 0
  BL, no; Week 3, yes; n=10 | 0
  BL, no; Week 3, no; n=10 | 10
  BL, yes; Week 4, yes; n=10 | 0
  BL, yes; Week 4, no; n=10 | 0
  BL, no; Week 4, yes; n=10 | 0
  BL, no; Week 4, no; n=10 | 10
  BL, yes; Week 5, yes; n=10 | 0
  BL, yes; Week 5, no; n=10 | 0
  BL, no; Week 5, yes; n=10 | 0
  BL, no; Week 5, no; n=10 | 10
  BL, yes; Week 6, yes; n=10 | 0
  BL, yes; Week 6, no; n=10 | 0
  BL, no; Week 6, yes; n=10 | 0
  BL, no; Week 6, no; n=10 | 10
  BL, yes; Week 7, yes; n=10 | 0
  BL, yes; Week 7, no; n=10 | 0
  BL, no; Week 7, yes; n=10 | 0
  BL, no; Week 7, no; n=10 | 10
  BL, yes; Week 8, yes; n=10 | 0
  BL, yes; Week 8, no; n=10 | 0
  BL, no; Week 8, yes; n=10 | 0
  BL, no; Week 8, no; n=10 | 10
  BL, yes; Week 12, yes; n=10 | 0
  BL, yes; Week 12, no; n=10 | 0
  BL, no; Week 12, yes; n=10 | 0
  BL, no; Week 12, no; n=10 | 10
  BL, yes; Week 16, yes; n=10 | 0
  BL, yes; Week 16, no; n=10 | 0
  BL, no; Week 16, yes; n=10 | 0
  BL, no; Week 16, no; n=10 | 10
  BL, yes; Week 20, yes; n=10 | 0
  BL, yes; Week 20, no; n=10 | 0
  BL, no; Week 20, yes; n=10 | 0
  BL, no; Week 20, no; n=10 | 10
  BL, yes; Week 24, yes; n=10 | 0
  BL, yes; Week 24, no; n=10 | 0
  BL, no; Week 24, yes; n=10 | 0
  BL, no; Week 24, no; n=10 | 10
  BL, yes; Week 28, yes; n=9 | 0
  BL, yes; Week 28, no; n=9 | 0
  BL, no; Week 28, yes; n=9 | 0
  BL, no; Week 28, no; n=9 | 9
  BL, yes; Week 36, yes; n=9 | 0
  BL, yes; Week 36, no; n=9 | 0
  BL, no; Week 36, yes; n=9 | 0
  BL, no; Week 36, no; n=9 | 9
  BL, yes; Week 48, yes; n=7 | 0
  BL, yes; Week 48, no; n=7 | 0
  BL, no; Week 48, yes; n=7 | 0
  BL, no; Week 48, no; n=7 | 7

28. Secondary Outcome: Mean Change From Baseline in the Immunoglobulin (Ig) Antibodies IgA, IgG, and IgM at Weeks 8, 24, and 48
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Low levels indicate immuno-suppression. IgA, IgG, and IgM were measured in the blood samples of the participants.
Time Frame: Baseline and Weeks 8, 24, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
g/L
  IgA, Week 8, n=9 | 0.014 (0.1337)
  IgA, Week 24, n=9 | -0.023 (0.0865)
  IgA, Week 48, n=7 | 0.086 (0.2889)
  IgG, Week 8, n=9 | 0.647 (0.9004)
  IgG, Week 24, n=10 | -0.150 (0.8641)
  IgG, Week 48, n=7 | -0.587 (0.9680)
  IgM, Week 8, n=7 | -0.063 (0.1482)
  IgM, Week 24, n=8 | -0.058 (0.1831)
  IgM, Week 48, n=5 | -0.108 (0.1809)

29. Secondary Outcome: Number of Participants Who Tested Positive/Negative for Human Anti-human Antibodies (HAHA) at Screening and at Weeks 24 and 48
Description: HAHA are indicators of immunogenicity to ofatumumab.
Time Frame: Screening; Weeks 24 and 48
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
participants
  Positive at Screening, n=10 | 0
  Negative at Screening, n=10 | 10
  Positive at Week 24, n=10 | 0
  Negative at Week 24, n=10 | 10
  Positive at Week 48, n=7 | 0
  Negative at Week 48, n=7 | 7

30. Secondary Outcome: Number of Participants With a Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: ECOG PS is used to assess how a participant's disease is progressing, to assess how the disease affects the daily living abilities of the participant, and to determine appropriate treatment and prognosis. The grades for the scale range from 0 (fully active) to 4 (completely disabled), with increasing severity.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 28, 36, and 48
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 10
participants
  Week 1, improved; n=10 | 0
  Week 1, deteriorated; n=10 | 0
  Week 2, improved; n=10 | 0
  Week 2, deteriorated; n=10 | 0
  Week 3, improved; n=10 | 0
  Week 3, deteriorated; n=10 | 0
  Week 4, improved; n=10 | 0
  Week 4, deteriorated; n=10 | 0
  Week 5, improved; n=10 | 0
  Week 5, deteriorated; n=10 | 0
  Week 6, improved; n=10 | 0
  Week 6, deteriorated; n=10 | 0
  Week 7, improved; n=10 | 0
  Week 7, deteriorated; n=10 | 0
  Week 8, improved; n=10 | 0
  Week 8, deteriorated; n=10 | 0
  Week 12, improved; n=10 | 0
  Week 12, deteriorated; n=10 | 0
  Week 16, improved; n=10 | 0
  Week 16, deteriorated; n=10 | 0
  Week 20, improved; n=10 | 0
  Week 20, deteriorated; n=10 | 0
  Week 24, improved; n=10 | 0
  Week 24, deteriorated; n=10 | 0
  Week 28, improved; n=9 | 0
  Week 28, deteriorated; n=9 | 0
  Week 36, improved; n=9 | 0
  Week 36, deteriorated; n=9 | 0
  Week 48, improved; n=7 | 0
  Week 48, deteriorated; n=7 | 0

31. Secondary Outcome: Maximum (Peak) Plasma Concentration (Cmax) of Ofatumumab
Description: Blood sampling on Day 1 and at Weeks 7 and 24 for pharmacokinetic (PK) evaluation was performed at the following time points: 0.5 hour (hr) before infusion; end of infusion; and 10 minutes (min), 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), and 120 hr (5 days) after infusion of ofatumumab. At Weeks 7 and 24, blood sampling was also performed 168 hr (7 days) and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Day 1; Weeks 7 and 24
Population: PK Parameter Population: all participants who received at least one dose of investigational drug, and in whom PK data were available and allowed parameter estimations. Only participants remaining in the study and contributing evaluable data at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per milliliter (mcg/mL)
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
Micrograms per milliliter (mcg/mL)
  Day 1, n=8 | 69.33 [43.15 to 111.39]
  Week 7, n=8 | 1670.36 [1324.95 to 2105.81]
  Week 24, n=7 | 864.93 [658.73 to 1135.69]

32. Secondary Outcome: Minimum Plasma Concentration (Cmin) of Ofatumumab
Description: Blood sampling at Weeks 7 and 24 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), 120 hr (5 days), 168 hr (7 days), and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Weeks 7 and 24
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
mcg/mL
  Week 7 | 832.17 [539.95 to 1282.55]
  Week 24 | 122.08 [28.75 to 518.37]

33. Secondary Outcome: Time to Reach Cmax (Tmax) Following Ofatumumab Administration
Description: Blood sampling on Day 1 and at Weeks 7 and 24 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), and 120 hr (5 days) after infusion of ofatumumab. At Weeks 7 and 24, blood sampling was also performed 168 hr (7 days) and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Day 1; Weeks 7 and 24
Population: PK Parameter Population. Only participants remaining in the study and contributing evaluable data at the indicated time points were analyzed.
Measure: Median (Full Range); unit: hr
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
hr
  Day 1, n=8 | 7.208 [6.00 to 16.50]
  Week 7, n=8 | 5.225 [4.47 to 6.30]
  Week 24, n=7 | 5.250 [4.00 to 28.65]

34. Secondary Outcome: Half-life (t1/2) of Ofatumumab
Description: t1/2 of ofatumumab is the time required for the plasma concentration of ofatumumab to decrease by half. Blood sampling on Day 1 and at Weeks 7 and 24 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), and 120 hr (5 days) after infusion of ofatumumab. At Weeks 7 and 24, blood sampling was also performed 168 hr (7 days) and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Day 1; Weeks 7 and 24
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
hr
  Day 1, n=8 | 9.585 [5.039 to 18.232]
  Week 7, n=8 | 331.275 [223.561 to 490.886]
  Week 24, n=7 | 300.354 [182.417 to 494.539]

35. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time t (AUC[0-t]) for Ofatumumab
Description: AUC(0-t) was evaluated from the plasma concentration versus time curve from time zero to the last measurable time point (time t). Blood sampling on Day 1 and at Weeks 7 and 24 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), and 120 hr (5 days) after infusion of ofatumumab. At Weeks 7 and 24, blood sampling was also performed 168 hr (7 days) and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Day 1; Weeks 7 and 24
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: hr*mcg/mL
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
hr*mcg/mL
  Day 1, n=8 | 1345.1 [466.0 to 3882.6]
  Week 7, n=8 | 587711.3 [332243.3 to 1039613.6]
  Week 24, n=7 | 283751.4 [106203.6 to 758118.2]

36. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 168 hr (AUC[0-168]) for Ofatumumab at Week 7
Description: Blood sampling at Week 7 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), 120 hr (5 days), 168 hr (7 days), and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Week 7
Population: PK Parameter Population
Measure: Geometric Mean (95% Confidence Interval); unit: hr*mcg/mL
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
hr*mcg/mL | 200181.8 [139285.0 to 287703.4]

37. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 672 hr (AUC[0-672]) for Ofatumumab at Week 24
Description: Blood sampling at Week 24 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), 120 hr (5 days), 168 hr (7 days), and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Week 24
Population: PK Parameter Population. Only participants contributing evaluable data at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*mcg/mL
Arm/Group | Ofatumumab
Number analyzed (Participants) | 7
hr*mcg/mL | 216678.1 [114237.9 to 410979.2]

38. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC[0-infinity]) for Ofatumumab
Description: as for outcome 33
Time Frame: Day 1; Weeks 7 and 24
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: hr*mcg/mL
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
hr*mcg/mL
  Day 1, n=8 | 1506.3 [594.0 to 3820.0]
  Week 7, n=8 | 716924.6 [374533.0 to 1372324.7]
  Week 24, n=7 | 302326.7 [122602.4 to 745511.3]

39. Secondary Outcome: Clearance (CL) of Ofatumumab From Plasma
Description: CL of ofatumumab from plasma of participants was evaluated. Blood sampling on Day 1 and at Weeks 7 and 24 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), and 120 hr (5 days) after infusion of ofatumumab. At Weeks 7 and 24, blood sampling was also performed 168 hr (7 days) and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Day 1; Weeks 7 and 24
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: mL/hr
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
mL/hr
  Day 1, n=8 | 199.157 [78.535 to 505.042]
  Week 7, n=8 | 9.991 [6.952 to 14.359]
  Week 24, n=7 | 9.230 [4.866 to 17.507]

40. Secondary Outcome: Volume of Distribution (Vz) During the Terminal Phase for Ofatumumab
Description: Vz for ofatumumab was calculated as a ratio of the amount of ofatumumab in the body during the terminal phase to the plasma concentration during the terminal phase. Blood sampling on Day 1 and at Weeks 7 and 24 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), and 120 hr (5 days) after infusion of ofatumumab. At Weeks 7 and 24, blood sampling was also performed 168 hr (7 days) and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Day 1; Weeks 7 and 24
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: mL
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
mL
  Day 1, n=8 | 2754.1 [1919.2 to 3952.2]
  Week 7, n=8 | 4774.9 [3610.7 to 6314.5]
  Week 24, n=7 | 3999.7 [2903.1 to 5510.4]

41. Secondary Outcome: Volume of Distribution at Steady State (Vss) for Ofatumumab
Description: Vss for ofatumumab was calculated as a ratio of the amount of ofatumumab in the body in equilibrium conditions to steady-state plasma concentrations. Blood sampling on Day 1 and at Weeks 7 and 24 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), and 120 hr (5 days) after infusion of ofatumumab. At Weeks 7 and 24, blood sampling was also performed 168 hr (7 days) and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Day 1; Weeks 7 and 24
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: mL
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
mL
  Day 1, n=8 | 3667.9 [2324.6 to 5787.5]
  Week 7, n=8 | 1333.8 [928.7 to 1915.4]
  Week 24, n=7 | 3069.2 [2122.9 to 4437.2]

42. Secondary Outcome: Mean Residence Time (MRTinf) of Ofatumumab
Description: MRTinf is the average amount of time that ofatumumab spends in the body. Blood sampling on Day 1 and at Weeks 7 and 24 for PK evaluation was performed at the following time points: 0.5 hr before infusion; end of infusion; and 10 min, 1 hr, 2 hr, 24 hr (1 day), 72 hr (3 days), and 120 hr (5 days) after infusion of ofatumumab. At Weeks 7 and 24, blood sampling was also performed 168 hr (7 days) and 336 hr (14 days) after infusion of ofatumumab.
Time Frame: Day 1; Weeks 7 and 24
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
hr
  Day 1, n=8 | 18.417 [10.437 to 32.500]
  Week 7, n=8 | 478.105 [333.067 to 686.300]
  Week 24, n=7 | 463.945 [263.535 to 816.762]

43. Other Pre Specified Outcome: Serum Hemolytic Complement Titer at Weeks 36 and 48: CH50
Description: The CH50 is the serum complement to lyse 50% of sensitized red blood cells; it's is a marker of complement activation. A high CH50 level suggests evidence for complement activation, whereas a low CH50 level suggests lack of complement activation.
Time Frame: Weeks 36 and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Kilo units per liter (KU/L)
Arm/Group | Ofatumumab
Number analyzed (Participants) | 8
Kilo units per liter (KU/L)
  Week 36, n=8 | 45.14 (13.643)
  Week 48, n=7 | 53.70 (11.818)

ADVERSE EVENTS:
Arm/Group | Ofatumumab
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=10)
Enteritis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=10)
Neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Blood lactate dehydrogenase increased (Investigations) | 5
Lymphocyte count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood glucose increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Protein total decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Weight increased (Investigations) | 1
Nasopharyngitis (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 4
Procedural complication (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis atrophic (Gastrointestinal disorders) | 1
Gingival swelling (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Influenza like illness (General disorders) | 1
Mucosal erosion (General disorders) | 1
Oedema peripheral (General disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Cataract (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Insomnia (Psychiatric disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.